CLINICAL TRIAL: NCT03486847
Title: Postoperative Atelectasis in Pediatric Patients With Prone Position : Effect of Repetitive Alveolar Recruitment by Lung Ultrasound
Brief Title: Postoperative Atelectasis in Pediatric Patients With Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-1802-088-923
Record Dates: First submitted 2018-03-26; First posted 2018-04-03 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Atelectasis, Postoperative; Atelectasis, Compression
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive recruitment with PEEP (Experimental): One alveolar recruitment at before surgery and repetitive alveolar recruitment (once an hour) during surgery
  Interventions: Procedure: Repetitive recruitment with PEEP
- One recruitment with PEEP (Active Comparator): One alveolar recruitment at before surgery
  Interventions: Procedure: One recruitment with PEEP

INTERVENTIONS:
Procedure: Repetitive recruitment with PEEP — Apply sustained airway pressure of 30-40 cmH2O for 10-20 seconds before suegery and once an hour during surgery. PEEP is set to 7 cmH2O.
  Arms: Repetitive recruitment with PEEP
Procedure: One recruitment with PEEP — Apply sustained airway pressure of 30-40 cmH2O for 10-20 seconds before surgery. PEEP is set to 7 cmH2O.
  Arms: One recruitment with PEEP

SUMMARY:
This study evaluates the incidence of postoperative atelectasis after general anesthesia with prone position using lung ultrasound in children age < 3 years.

DETAILED DESCRIPTION:
Atelectasis is common in pediatric patients after general anesthesia. Particularly, infants are more likely to develop atelectasis or ventilation-perfusion imbalance after general anesthesia because of the immature ribs and respiratory muscles, the high compliance of the rib cage and a significant reduction in functional residual capacity (FRC) during general anesthesia. Previous studies have reported that alveolar recruitment and positive end-expiratory pressure (PEEP) can be used to reduce atelectasis in children. Also, previous studies have shown that the lung ultrasound can be used to evaluate the degree of atelectasis during general anesthesia in children.

However, none of the previous studies investigated the incidence of atelectasis, the effect of alveolar recruitment, and the PEEP in pediatric patients under general anesthesia with prone position. The purpose of this study was to evaluate previously described parameters using lung ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing general anesthesia with prone position
* Endotracheal intubation and mechanical ventilation during general anesthesia
* Operation time is more than 2 hours

Exclusion Criteria:

* Previous lung surgery
* Any abnormal findings such as atelectasis, pneumothorax, pleural effusion, or pneumonia on preoperative chest X-ray
* Researchers judge (to be inappropriate)

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of pre-extubation atelectasis | postoperative 10 minutes
  Incidence of pre-extubation atelectasis accessed by lung ultrasound

SECONDARY OUTCOMES:
Incidence of intraoperative atelectasis after intubation | intraoperative
  Incidence of intraoperative atelectasis after induction accessed by lung ultrasound
Incidence of intraoperative atelectasis after position change to prone | intraoperative
  Incidence of intraoperative atelectasis after position change to prone accessed by lung ultrasound
Incidence of intraoperative and postoperative (within 12hr) desaturation | intraoperative and postoperative (within 12hr)
  Oxygen saturation by pulse oximetry (SpO2) ≤ 95% or 10% below the baseline value
Incidence of intraoperative hypotension | intraoperative
  Systolic blood pressure (SBP) ≤ 20% below the baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Hee Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongnogu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jang YE, Ji SH, Kim EH, Lee JH, Kim JT, Kim HS. Effect of regular alveolar recruitment on intraoperative atelectasis in paediatric patients ventilated in the prone position: a randomised controlled trial. Br J Anaesth. 2020 May;124(5):648-655. doi: 10.1016/j.bja.2020.01.022. Epub 2020 Mar 10. PMID 32169254